CLINICAL TRIAL: NCT00667199
Title: A Double Blind, Dose Response Phase II, Multicentre Study of Radium 223 (Alpharadin®) for the Palliation of Painful Bone Metastases in Hormone Refractory Prostate Cancer Patients
Brief Title: BAY88-8223, Does Response Study in HRPC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15305; BC1-03 (Other: Algeta ASA); 2004-000299-15 (EudraCT Number)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Hormone Refractory Prostate Cancer; Bone Metastases
Keywords: Hormone Refractory Prostate Cancer; Bone Metastases; Radium-223; Palliation of bone pain
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Radium-223 dichloride (Xofigo, BAY88-8223)-5kBq/kg (Experimental): Each patient received a single injection of radium-223 , based on the randomised dose level (5kBq/kg) and individual body weight.
  A second injection of radium-223 set to 50 kBq/kg b.w. could be offered to patients in the Follow-up Period at the discretion of the investigator.
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)
- Radium-223 dichloride (Xofigo, BAY88-8223)-25 kBq/kg (Experimental): Each patient received a single injection of radium-223 , based on the randomised dose level (25kBq/kg) and individual body weight.
  A second injection of radium-223 set to 50 kBq/kg b.w. could be offered to patients in the Follow-up Period at the discretion of the investigator.
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)
- Radium-223 dichloride (Xofigo, BAY88-8223)-50 kBq/kg (Experimental): Each patient received a single injection of radium-223 , based on the randomised dose level (50kBq/kg) and individual body weight.
  A second injection of radium-223 set to 50 kBq/kg b.w. could be offered to patients in the Follow-up Period at the discretion of the investigator.
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)
- Radium-223 dichloride (Xofigo, BAY88-8223)-100 kBq/kg (Experimental): Each patient received a single injection of radium-223 , based on the randomised dose level (100kBq/kg) and individual body weight.
  A second injection of radium-223 set to 50 kBq/kg b.w. could be offered to patients in the Follow-up Period at the discretion of the investigator.
  Interventions: Drug: Radium-223 dichloride (BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (BAY88-8223) — The required volume of study drug to be administered to a patient was calculated using the patient's body weight, the dose (5 , 25 , 50 or 100 kBq/kg b.w.)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the investigational radioisotope Radium-223, Xofigo (Alpharadin), in treatment of men with prostate cancer and bone metastases that no longer respond to hormonal treatment.

DETAILED DESCRIPTION:
The study is designed to investigate whether there is a dose-response relationship for radium-223 in patients with painful bone metastases secondary to prostate carcinoma regarding palliation of bone pain. The palliative efficacy will be established through assessments of bone pain and consumption of analgesia. Furthermore, the aim is to find the most efficient dose with an acceptable safety profile. The safety will be assessed through measurements of adverse events, and acute haematological toxicity during the study period. Long-term chronic toxicity, and the overall survival at one and two years post treatment will also be assessed.

This is a double-blind, dose-response, randomized, multi-centre phase II efficacy and safety study of radium- 223. The clinical sites will enroll a total of 100 eligible patients. The treatment is a single intravenous administration of radium-223.

The target population is patients suffering from bone pain due to skeletal metastasis secondary to hormone refractory prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* Histologically/cytologically confirmed adenocarcinoma of the prostate
* Patient is hormone refractory with evidence of progressive disease:

  * Patient must be maintained on androgen ablation therapy with LHRH agonist or have undergone orchiectomy
  * Patient's testosterone level is required to be equal to or below 50 ng/dl
  * Patients in which flutamide, nilutamide, megestrol acetate, polyestradiol phosphate, aminoglutethimide, and ketoconazole, has been recently withdrawn must demonstrate progression of disease and be at last 4 weeks beyond the discontinuation of such agents; for bicalutamide 6 weeks is required
  * Increase in PSA levels in two consecutive measurements with at least one week apart, demonstrating an increase over the reference (nadir) value, and with the final PSA >/= 5 ng/ml

    * A reference PSA (nadir) value must be measured at least 4 weeks after the discontinuation of flutamide, nilutamide, megestrol acetate, polyestradiol phosphate, aminoglutethimide, and ketoconazole, and at least 6 weeks after discontinuation of bicalutamide
    * If the third PSA value is lower than the second value, the patient could still be eligible, provided a fourth measurement obtained at least 1 week after the third PSA value, is grater than the second PSA value and >/= 5 ng/ml
* Multifocal (>1) skeletal metastases confirmed by bone scintigraphy within 6 weeks
* Bone pain with a score of at least 2 on BPI average pain, despite adequate use of analgesics, that correlates with areas of increased uptake (osteoblastic activity) on bone scintigraphy
* Performance status: ECOG 0-2 or Karnofsky >/= 60%
* Life expectancy: At least 3 months
* Age more than 40 years
* Laboratory requirements:

  * Neutrophil count >/= 1,5 x 109/L
  * Platelet count >/= 100 x109/L
  * Hemoglobin > 95 g/L
  * Bilirubin within normal institutional limits
  * ASAT and ALAT <2,5 times upper limit of normal (ULN)
* The patient is willing and able to comply with the protocol (including maintenance of patient diary, completion of pain assessment forms), and agrees to return to the hospital for follow-up visits and examinations
* The patient has been fully informed about the study and has signed the informed consent form

Exclusion criteria

* Has received an investigational drug within 4 weeks before the administration of radium-223, or is scheduled to receiving one during the study period
* Has received chemo-, immunotherapy, or external radiotherapy within the last 4 weeks prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Has received prior hemibody external radiotherapy
* Has received systemic radiotherapy with strontium-89, samarium-153, rhenium-186 or rhenium 188 for the treatment of bony metastases within the last year prior to inclusion
* Has started treatment with bisphosphonates less than 3 months prior to administration of study drug
* Patients experiencing hormone withdrawal syndrome, or are </= 4 weeks post withdrawal of antiandrogen therapy (6 weeks for bicalutamide)
* Patients who have started steroids or changed to treatment with steroids within the last 4 weeks prior to administration of radium-223
* Has other clinically significant or symptomatic disease, which might interfere with the assessment of bone pain, e.g. spinal cord compression, compression or infiltration of a neural plexus, nerve root or peripheral nerves
* Other currently active (relapse within the last 3 year) malignancy (except non-melanoma skin cancer), or known brain or visceral metastases dominating the clinical picture of the patient
* Other serious illness or medical condition:

  * any uncontrolled infection
  * cardiac failure Classification III or IV (New York Heart Association)
  * Crohn disease or Ulcerative colitis
  * known bone fracture within 8 weeks

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-05-30 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2009-10-06 (Actual)

PRIMARY OUTCOMES:
Pain Assessment (using a 100mm Visual Analogue Scale) | 16 weeks
Analgesic consumption | 16 weeks

SECONDARY OUTCOMES:
Reduction of pain: the pain dimension of Quality of Life assessed using the Brief Pain Inventory (BPI) form, with total pain score and subtotals, after injection and compared to scores at baseline | 16 weeks
Duration of pain relief: measured as the time between the first and last evaluation time points at which the pain response criteria were met | 16 weeks
The safety of radium-223: the total safety profile including adverse events and clinical laboratory measurements, with emphasis on haematological toxicity. Adverse events will be recorded continuously during the study period. | 2 years
The date of death (if within 24 months after the injection of study drug) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- [Result] Nilsson S, Strang P, Aksnes AK, Franzen L, Olivier P, Pecking A, Staffurth J, Vasanthan S, Andersson C, Bruland OS. A randomized, dose-response, multicenter phase II study of radium-223 chloride for the palliation of painful bone metastases in patients with castration-resistant prostate cancer. Eur J Cancer. 2012 Mar;48(5):678-86. doi: 10.1016/j.ejca.2011.12.023. Epub 2012 Feb 15. PMID 22341993